CLINICAL TRIAL: NCT07010406
Title: A Phase 1, Open-label, Randomized, 2-part Study to Evaluate the Relative Bioavailability of Povetacicept Formulations and Bioequivalence of Povetacicept Presentations in Healthy Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability of Povetacicept Formulations and Bioequivalence of Povetacicept Presentations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX24-AIS-D11
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A1: Povetacicept Bioavailability (Experimental): Participants will be randomized to receive one of the two Povetacicept formulations.
  Interventions: Drug: Povetacicept
- Part A2: Povetacicept Bioavailability (Experimental): Participants will be randomized to receive one of the two Povetacicept formulations.
  Interventions: Drug: Povetacicept
- Part B1: Povetacicept Bioequivalence (Experimental): Participants will be randomized to receive one of the two Povetacicept presentations.
  Interventions: Drug: Povetacicept
- Part B2: Povetacicept Bioequivalence (Experimental): Participants will be randomized to receive one of the two Povetacicept presentations.
  Interventions: Drug: Povetacicept

INTERVENTIONS:
Drug: Povetacicept — Injection for Subcutaneous Administration.

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of Povetacicept formulations, bioequivalence of Povetacicept presentations, and safety and tolerability of Povetacicept.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2), inclusive
* A total body weight of more than (>) 50 kg

Key Exclusion Criteria:

* History of febrile illness that has not fully resolved within 14 days before the dose of study drug.
* Immunization with a live vaccine within 45 days before study drug administration or a non live vaccine within 14 days before study drug administration.

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve From the Time of Dosing to 28 Days (AUC0-28d) of Free Povetacicept | From Day 1 up to Day 30
Maximum Observed Plasma Concentration (Cmax) of Free Povetacicept | From Day 1 up to Day 30

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 31

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Celerion - Tempe, Tempe, Arizona
  - Celerion - Lincoln, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing